CLINICAL TRIAL: NCT00239057
Title: Enteric-Coated Mycophenolate Sodium (EC-MPS) Administration in Maintenance Renal Transplant Patients Receiving Cyclosporine Microemulsion (CsA-ME) and Steroids, for the Withdrawal of Concomitant Steroid Therapy: a Prospective, Open-label, Exploratory Study
Brief Title: Study of Enteric-coated Mycophenolate Sodium Maintenance Therapy in Patients With Renal Transplant Receiving Cyclosporine Microemulsion and Steroids,
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405IT03
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Maintenance Renal Transplantation
Keywords: Renal transplantation, EC-MPS

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium

SUMMARY:
The aim of this study is to evaluate if the addition of EC-MPS to CsA-ME allows the safe withdrawal of the concomitant corticosteroid therapy in long-term maintenance renal allograft recipients.

All patients of the core study who are interested of being treated with EC-MPS will be included in an open-label extension study to collect further information on the long-term safety, tolerability and efficacy of this drug.

ELIGIBILITY:
Inclusion criteria

1. Male or female, 18 years of age or older. 2. Recipients of first or secondary cadaver, living related or unrelated donor kidney transplant performed at least 6 month before screening (Visit 1) 3. Patients currently receiving CsA-ME and corticosteroids (at least 5 mg of prednisone equivalents) for at least 3 months prior to Screening, with or without Mycophenolate mofetil or azathioprine.

4. Serum creatinine levels < 2.3 mg/dL (=204 µmol/L) at screening and at baseline 5. Stable kidney function, i.e. increase in serum creatinine less than 20% in the last 3 months before screening and at baseline (baseline value as compared to the value obtained at screening) Exclusion Criteria

1. Multi-organ recipients (e.g., kidney and pancreas, double kidneys) or previous transplant with any other organ different from kidney
2. Patients whit a second transplant who rejected the first one for immunological reasons or because of the relapse of the autoimmune disease which leaded to the end-stage renal failure
3. Histological evidence of acute rejection or treatment for acute rejection within the three months prior to Screening, or histological signs or clinical signs of chronic rejection (as significant proteinuria, i.e. > 300 mg/24 hours.
4. Patients with maintenance steroid therapy for other diseases (i.e. autoimmune diseases, Lupus).
5. Patients with any known hypersensitivity to EC-MPS or other components of the formulation (e.g., lactose)
6. Patients with thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<4,000/mm3), and/or anemia (hemoglobin <9.0 g/dL) prior to Screening visit.
7. Patients who have received an investigational drug within two weeks prior to Screening visit.
8. Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
9. Females of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, who are unwilling to use effective means of contraception
10. Presence of clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus that would interfere with the appropriate conduct of the study.
11. Any changes of immunosuppressive regimen due to graft malfunction, or any known clinically significant physical and/or laboratory changes in the 2 months prior to Screening visit.
12. Known positivity for HIV, HBsAg
13. Active viral hepatitis, as shown by liver function tests (AST or ALT) higher than twice the upper limit of normality
14. Evidence of drug and/or alcohol abuse Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-05; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy prove acute rejection requiring treatment within six months of the start of the study.

SECONDARY OUTCOMES:
Assessment of the changes in body-weight, blood pressure, serum lipid levels, renal function, glaciated hemoglobin, dermatological condition and quality of life six months after the start of the study
Safety and tolerability
Pharmacokinetics of MPA and MPAG in the patient subgroup that was receiving MMF (screening period) before the start of the study and two weeks after the start of the administration of EC-MPS.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis